CLINICAL TRIAL: NCT02051049
Title: Long-term Safety Follow-up Study of Patients Having Received Infusions of HepaStem
Brief Title: Long-term Safety Follow-up Study of Patients Having Received HepaStem (SAF001)
Status: Completed | Type: Observational
Sponsor: Cellaion SA (Industry)
Responsible Party: Sponsor
Other Study IDs: SAF001
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Urea Cycle Disorders; Crigler Najjar Syndrome
Keywords: CN; UCD
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Crigler-Najjar Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Inborn errors of liver metabolism

SUMMARY:
The purpose of this study is to assess the long-term safety follow-up of patients having been treated with HepaStem.

DETAILED DESCRIPTION:
The primary objective of the SAF001 study is the long-term safety surveillance of the patients post infusion with HepaStem. Furthermore, the evolution of both the metabolic condition and the quality of life are followed. As much as possible, the surveillance will mimic the standard follow-up of the respective diseases (standard of care). The surveillance will end when the patient is undergoing an organ transplant or takes part in another research study. This surveillance will last up to a maximum of 48 months.

ELIGIBILITY:
Main Inclusion Criteria:

- Subject having received HepaStem during a former interventional clinical study and who have terminated their participation in that study.

Exclusion Criteria:

- Subject has received mature liver cells, stem cells transplantation other than HepaStem, or organ liver transplant.

Max Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The SAF001 study will include all patients having received infusions of HepaStem in any former interventional study conducted by Promethera Biosciences.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-03; Primary Completion 2018-04 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Characterisation of the long term safety profile of HepaStem therapy. | 4 years
  Assessment of safety will be achieved by evaluating the following parameters
  * Physical examination
  * Vital signs
  * Laboratory tests
  * Liver tumor markers
  * Autoimmune markers related to liver pathology
  * Anti-HLA antibodies specific for donor cell haplotypes
  * Morphology of liver, bile ducts, and portal system by ultrasound
  * Morphology of the kidneys by ultrasound
  * Non-serious or serious Adverse Events of Special Interest (AESIs) and Serious Adverse Events (SAEs) related to HepaStem therapy.

SECONDARY OUTCOMES:
To characterize the disease evolution after having received HepaStem therapy and to report on general safety. | 4 years
  This assessment is based on the evaluation of:
  * Report on cognitive skills, behaviour, and health-related quality of life indicators
  * Non-serious or serious Adverse Events of Special Interest (AESIs) and Serious Adverse Events (SAEs) related to concomitant medications or other causes
  Indication I: Crigler-Najjar syndrome
  * Frequency and severity of metabolic decompensation
  * Metabolic parameters (serum total bilirubin)
  * Report on supportive treatment and any adjustment of phototherapy and medication (eg phenobarbital treatment)
  Indication II: Urea cycle disorders
  * Frequency and severity of metabolic decompensation
  * Metabolic parameters (NH3 values, amino acids in plasma)
  * Report on supportive treatment and any adjustment of:
    * diet (natural protein intake, total protein intake, amino acid supplements)
    * Medication (eg nitrogen scavengers)

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Smets, MD, Principal Investigator — Cliniques universitaires Saint-Luc (Belgium); Dries Dobbelaere, MD/Prof, Principal Investigator — CHRU de Lille - Hopital Jeanne de Flandre (France); Isabel Gonçalves, MD/Prof, Principal Investigator — Hospital Pediátrico de Coimbra (Portugal); Stephanie Grunewald, MD, Principal Investigator — Great Ormond Street Children Hospital; Giuliano Torre, MD, Principal Investigator — IRCCS OSPEDALE PEDIATRICO DEL BAMBINO GESÃ (Roma); Hanna Mandel, MD, Principal Investigator — Rambam Health Corporation
Locations (1):
- Promethera Biosciences, Mont-Saint-Guibert, Belgium